CLINICAL TRIAL: NCT03253562
Title: Comparative Efficacy and Safety of Vildagliptin Versus Metformin in Reduction of Cardiovascular Complications in Type 2 Diabetic Patients With Hypertension
Brief Title: Metformin Versus Vildagliptin for Diabetic Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Dalia Kamal Zaafar Ali, assistant lecturer of pharmacology and toxicology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE00217
Record Dates: First submitted 2017-08-10; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Reducing the Elevated Blood Pressure for Diabetic Hypertensive Patients
Keywords: diabetes; Metformin; vildagliptin; hypertension; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Metformin; Vildagliptin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy control (No Intervention): healthy volunteers not suffering from diabetes or hypertension
- diabetic hypertensive recently diagnosed patients (No Intervention): recently diagnosed patients suffers from diabetes type 2 and hypertension but didnot receive their proper treatment yet
- Metformin treated group (Other): diabetic hypertensive patients which were treated with captopril for their hypertension and metformin for their diabetes
  Interventions: Drug: Metformin Pill
- Vildagliptin treated group (Other): diabetic hypertensive patients which were treated with captopril for their hypertension and vildagliptin for their diabetes
  Interventions: Drug: Vildagliptin 50 mg

INTERVENTIONS:
Drug: Metformin Pill — a biguanide used as an insulin sensitizer for patients suffering from type 2 diabetes mellitus
  Arms: Metformin treated group
Drug: Vildagliptin 50 mg — Dpp4i antihyperglycemic drug used for treatment of type 2 diabetes mellitus
  Arms: Vildagliptin treated group

SUMMARY:
This is a controlled study to measure the efficacy of using metformin or vildagliptin for type 2 diabetic patients who suffers from hypertension to reduce cardiovascular risk resulting from both diabetes and hypertension using different parameters measuring

DETAILED DESCRIPTION:
Several studies indicated that type 2 diabetes mellitus and hypertension are associated with increased cardiovascular complications. Recently, studies suggest that metformin and vildagliptin can reduce cardiovascular complications in diabetic patients with unclear mechanisms. This work aimed to determine the effect of metformin and vildagliptin on diabetic-hypertensive patients. Patients were allocated into four groups: groupI: healthy volunteers, groupII: patients recently diagnosed with their hypertension and diabetes, groupIII: patients treated with captopril (25mg once daily) for their hypertension in addition to metformin (1000mg bid) groupIV: patients treated with captopril (25mg bid) for hypertension in addition to vildagliptin (50mg bid). At the end of the therapeutic period, then total cholesterol, LDL,serum Creatinine level, blood pressure and vascular endothelial growth factor (VEGF) levels in serum will be measured for different groups to estimate the benefits of one drug over the other one in protecting against cardiovascular risks for diabetic hypertensive patients..

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from moderate HTN and DM, their HbA1c ≥ 7 and age range between 40-60 years, treatment with diet alone, any combination of oral antidiabetic agents and/or insulin before admission

Exclusion Criteria:

* Clinical evidence of ischemic heart disease, chronic obstructive pulmonary disease, presence of diabetic ketoacidosis (DKA), patients admitted to intensive care unit (ICU), subjects expected to undergo surgery during the study period, patients with clinically relevant hepatic disease, impaired renal function (serum creatinine ≥3.0 mg/dL), systemic infections or pregnancy. Also, patients on medications known to interfere with the blood glucose level (either increasing or decreasing) were excluded from the study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
benefit of reducing hypertension in diabetic hypertensive patients | 6 months
  blood pressure will be measured
benefit of lowering cardiovascular risks for diabetic hypertensive patients | 6 months
  total lipid profile will be measured
benefit of improving the condition of elevated blood pressure in patients through neovascularization | 6 months
  vascular endothelial growth factor level in serum will be measured

SECONDARY OUTCOMES:
reducing obesity for diabetic patients | 6months
  difference in body weight at the beginning and the end of the study will be measured
comparing the anti-hyperglycemic effect of each drug for diabetic hypertensive patients | 6 months
  glycated hemoglobin will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Hekma A Abdel-Latif, Professor, Study Chair — cairo university faculty of pharmacy; Abdel Rahman M El-Naggar, Professor, Study Director — Cairo University; Mohammed F Elyamany, assistant professor, Study Director — cairo university faculty of pharmacy; Soha O Hassanin, lecturer, Study Director — MTI unuversity faculty of pharmacy; Atef Bassyouni, Professor, Study Director — National institute of diabetes and endocrinology; Dalia K Zaafar, assistant lecturer, Principal Investigator — MTI unuversity faculty of pharmacy
Locations (1):
- National institute of diabetes and endocrinology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No